CLINICAL TRIAL: NCT00246116
Title: Functional Imaging of Treatment Effects: A Companion Protocol to a Phase II Study of Extracranial Stereotactic Radioablation (a.k.a. Stereotactic Body Radiotherapy) in Early Stage Non-Small Cell Lung Cancer.
Brief Title: Functional Imaging of Treatment Effects: A Companion Protocol to a Study of Extracranial Stereotactic Radioablation in Early Stage Non-Small Cell Lung Cancer
Acronym: SBF Companion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0201-06
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Non-small-cell Lung Cancer
Keywords: Lung Cancer; Radiation Oncology; Treated with Stereostatic Body Radiation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Functional Imaging of Treatment Effects — PET & VQ Scans

SUMMARY:
For this companion protocol, we intend to make an assessment of both tumor response and local tissue effects. Patients undergoing the correlative investigation will be a subset of the patients already enrolled on the phase II study.

DETAILED DESCRIPTION:
One of the shortcomings of the trial design recognized in the phase I study had to do with the assessment of local effects, both relating to tumor control and adjacent tissue toxicity. For example, response rates were generally incomplete to the therapy, especially at the lower dose level cohorts, and it was not clear if those patients had residual viable tumor capable of sustaining growth. Repeat biopsies in this population are prohibitively toxic. We generally followed these patients with chest x-rays and CT's until there was evidence of progression. At that point, we would perform a PET scan and repeat systemic staging. Since the majority of patients will retain residual "abnormalities" worrisome for residual disease, ideally, there would be data or testing capable of characterizing these abnormalities earlier in the post-treatment course. In the same token, several patients in the phase I study had post treatment imaging changes around the tumor targets. If these patients had symptomatic decline, it was never clear if the treatment effects around the target were actually involved in the overall decline. Certainly, the patient population selected has other medical problems that will continue to cause poor health. Ideally, though, we would refer to data indicating the degree of damage to surrounding normal lung from the ESR such that a realistic assessment of percentage of overall organ damage from the therapy can be ascertained.

ELIGIBILITY:
Inclusion Criteria:

* Patients consented, eligible, and scheduled to be treated on the phase II study of extracranial stereotactic radioablation (a.k.a stereotactic body radiotherapy) for early stage lung cancer already approved at Indiana University

Exclusion Criteria:

* Patients with contraindications to functional imaging (e.g. allergy to agent used in studies) and patient unwilling to fulfill requirements of both protocols are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2002-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To characterize the effect of treatment on tumor metabolic activity as a function of time. | 5 years from enrollment

SECONDARY OUTCOMES:
To correlate the first two objectives with outcome objectives of the clinical phase II protocol (survival, local control, and toxicity) in order to assess the ultimate utility of these imaging assessments in this patient population. | 5 years from completion of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Ronald McGarry, MD, Principal Investigator — Indiana University - Department of Radiation Oncology

REFERENCES:
- See also: Link to Department of Radiation Oncology — http://www.medicine.iu.edu/body.cfm?id=4491